CLINICAL TRIAL: NCT00716456
Title: A Phase I/II Trial of Cetuximab in Patients With Lung Adenocarcinoma Receiving Erlotinib That Have Developed "Acquired Resistance" to Erlotinib
Brief Title: Cetuximab in Patients With Lung Adenocarcinoma Receiving Erlotinib That Have Developed "Acquired Resistance" to Erlotinib
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-055
Record Dates: First submitted 2008-07-15; First posted 2008-07-16 (Estimated); Results first posted 2015-04-30 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Lung Adenocarcinoma
Keywords: MAB C225(CETUXIMAB)(ANTI-EGFR); OSI-774, TARCEVA (ERLOTINIB); Lung; Adenocarcinoma; Lung cancer
MeSH Terms: conditions — Adenocarcinoma of Lung; Adenocarcinoma; Lung Neoplasms | interventions — Erlotinib Hydrochloride; Cetuximab

ARMS (1):
- 1 (Experimental): In the phase I portion, patients will be enrolled in cohorts of 3-6 patients;receiving daily erlotinib 100 mg along with cetuximab given every 2 weeks beginning at 250mg/m2 IV. Following the initial dose, for dose levels 1 and 2 (250 mg/m2 and 375 mg/m2) patients will receive treatment every 2 weeks with cetuximab over 60 minutes. For dose level 3 (500 mg/m2) patients will receive treatment every 2 weeks with cetuximab over 120 minutes. The infusion rate of cetuximab should never exceed 10 mg/minute (5 mL/min). The dose may subsequently be reduced for individual patients, depending on a patient's toxicity.
  Interventions: Drug: erlotinib with cetuximab

INTERVENTIONS:
Drug: erlotinib with cetuximab — The phase I portion will accrue as many as 3 cohorts of 3-6 patients; receiving erlotinib 100 mg daily along with escalating doses of cetuximab administered every 2 weeks beginning at 250mg/m2 IV without a loading dose. Subsequent cetuximab dose levels will be 375 mg/m2, and 500 mg/m2, administered IV every 2 weeks. Patients will have baseline CT, labs and ECG done within 2 weeks of study entry. Three patients will be enrolled per dose level. Patients will be monitored for toxicity weekly for the first 5 weeks, and every 2 weeks thereafter. Patients will be monitored for response by CT in the fourth week of combined therapy and every 8 weeks. All patients in this portion of the trial will receive intravenous cetuximab every two weeks at the MTD (to be determined in phase I portion) and daily erlotinib on an outpatient basis and will obtain clinical re-evaluation and radiographic re-imaging on a schedule similar to that followed in the phase I portion

SUMMARY:
The purpose of this study is to test if cetuximab (Erbitux) can shrink lung cancers that initially became smaller after taking erlotinib and then started to get bigger despite continuing treatment. Cetuximab is a medicine approved by the U.S. Food and Drug administration for treatment of head and neck and colon cancer. The goal of the phase I portion of this trial is to find out the highest dose of cetuximab that can be taken together with erlotinib. This study will also give an idea of how well cetuximab shrinks lung cancer when given with erlotinib.

The purpose of this study is to test if cetuximab (Erbitux) can shrink lung cancers that initially became smaller after taking erlotinib or gefitinib and then started to get bigger despite continuing treatment. Cetuximab is a medicine approved by the U.S. Food and Drug administration for treatment of head and neck and colon cancer. The goal of this phase is to determine if cetuximab given with erlotinib causes lung cancers to shrink in size.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic evidence of lung adenocarcinoma confirmed at MSKCC
* Measurable (RECIST) indicator lesions not previously irradiated
* Radiographic progression by RECIST during treatment with erlotinib
* Received treatment with erlotinib throughout the one month prior to enrollment
* Received treatment with erlotinib for >3 months
* At least one of the following:
* Previously received treatment with erlotinib, gefitinib, or an investigational EGFR TK inhibitor (patients may have received other treatments subsequently including radiation or chemotherapy) and had a radiographic partial or complete response to treatment as defined by RECIST criteria
* A documented mutation in EGFR exons 19 or 21.
* Karnofsky performance status ≥ or = to 70%
* Total bilirubin: within normal institutional limits. AST/(SGOT)/ALT(SGPT)< or = to 2.5 X institutional upper limit of normal (ULN)
* Signed informed consent
* Effective contraception *
* Age > 18 years old *Sexually active women of childbearing potential must use an effective method of birth control during the course of the study, in a manner such that risk of failure is minimized. Prior to study enrollment, women of childbearing potential (WOCBP) must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy. In addition, men enrolled on this study should understand the risks to any sexual partner of childbearing potential and should practice an effective method of birth control. All WOCBP MUST have a negative pregnancy test within two weeks prior to first receiving investigational product. If the pregnancy test is positive, the patient must not receive investigational product and must not be enrolled in the study. In addition, all WOCBP should be instructed to contact the Investigator immediately if they suspect they might be pregnant (e.g., missed or late menstrual period) at any time during study participation. The Investigator must immediately notify BMS in the event of a confirmed pregnancy in a patient participating in the study.

Exclusion Criteria:

* CNS lesions which are symptomatic and/or requiring escalating doses of corticosteroids.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Prior cetuximab or panitumumab. Prior severe infusion reaction to a monoclonal antibody.
* Current grade 2 or greater skin toxicity on erlotinib therapy
* Radiotherapy ≤ or = to 14 days prior to enrollment
* Any investigational agent or therapy ≤ or = to 30 days before enrollment
* Systemic chemotherapy, hormonal therapy, immunotherapy, or experimental or approved proteins/antibodies (except erlotinib) ≤ or = to 30 days before enrollment
* Women who are pregnant or lactating.
* Known positive test(s) for human immunodeficiency virus infection, hepatitis C virus, acute or chronic active hepatitis B infection
* Major surgery within 28 days or minor surgery within 14 days of study enrollment
* Men or women of child-bearing potential (women who are post-menopausal < 52 weeks, not surgically sterilized, or not abstinent) not consenting to use adequate contraception (per institutional standard of care) during the course of the study and after the last investigational product(s) administration (24 weeks for women, 4 weeks for men)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2008-07; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Riely, PhD, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memoral Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan-Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center at Mercy Medical Center, Rockville Centre, New York
  - Memoral Sloan Kettering Cancer Center at Phelps, Sleepy Hollow, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol Open to Accrual: 7/15/2008
  Protocol Closed to Accrual: 5/25/2010
  Primary Completion Date: 5/24/2011
  Recruitment Location is the Medical Clinic
Groups:
- Cetuximab 250 mg/m2: Cetuximab 250 mg/m2 IV every two weeks
- Cetuximab 375 mg/m2: Cetuximab 375 mg/m2 IV every two weeks
- Cetuximab 500 mg/m2: Cetuximab 500 mg/m2 IV every two weeks
Period: Overall Study
Arm/Group | Cetuximab 250 mg/m2 | Cetuximab 375 mg/m2 | Cetuximab 500 mg/m2
Started | 3 | 5 | 13
Completed | 3 | 3 | 13
Not Completed | 0 | 2 | 0
Not completed — Adverse Event | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cetuximab 250 mg/m2 | Cetuximab 375 mg/m2 | Cetuximab 500 mg/m2 | Total
Number analyzed (Participants) | 3 | 5 | 13 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 9 | 12
  >=65 years | 2 | 3 | 4 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 9 | 14
  Male | 2 | 1 | 4 | 7
Region of Enrollment [Number; unit: participants]
  United States | 3 | 5 | 13 | 21

OUTCOME MEASURES:

1. Primary Outcome: The Maximum Tolerated Dose (MTD) of Cetuximab Given Every 2 Weeks
Description: To determine the maximum tolerated dose (MTD) of cetuximab given every 2 weeks in patients with lung adenocarcinoma receiving erlotinib that have developed acquired resistance to erlotinib (phase I portion)
Time Frame: At conclusion of study, up to 24 weeks
Measure: Number; unit: mg/m2 of CETUXIMAB
Arm/Group | Cetuximab 250 mg/m2 | Cetuximab 375 mg/m2 | Cetuximab 500 mg/m2
Number analyzed (Participants) | 3 | 5 | 13
mg/m2 of CETUXIMAB | 500 | 500 | 500

ADVERSE EVENTS:
Arm/Group | Cetuximab 250 mg/m2 | Cetuximab 375 mg/m2 | Cetuximab 500 mg/m2
Serious Adverse Events (participants affected / at risk) | 3/3 | 2/5 | 5/13
Other Adverse Events (participants affected / at risk) | 3/3 | 3/5 | 12/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cetuximab 250 mg/m2 (N=3) | Cetuximab 375 mg/m2 (N=5) | Cetuximab 500 mg/m2 (N=13)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Allergic reaction/Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Renal Failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase (Investigations) | 0 (0) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cetuximab 250 mg/m2 (N=3) | Cetuximab 375 mg/m2 (N=5) | Cetuximab 500 mg/m2 (N=13)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (2) | 7 (15)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Fatigue (General disorders) | 2 (8) | 3 (3) | 5 (9)
Fever (General disorders) | 1 (1) | 1 (2) | 3 (3)
Hemorrhage, Nose (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Inf unknown ANC-Ungual (Nails) (Infections and infestations) | 0 (0) | 2 (4) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 2 (6) | 4 (27)
Mucositis-Oral (Gastrointestinal disorders) | 1 (1) | 2 (2) | 4 (8)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 7 (10)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (5) | 2 (2)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (15) | 11 (17)
Rash acne/acneiform (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes